CLINICAL TRIAL: NCT02525731
Title: Collaborative Care Intervention to Improve Providers' Opioid Prescribing for HIV-infected Patients - Patient Cohort Component
Brief Title: Targeting Effective Analgesia in Clinics for HIV - Patient Cohort
Acronym: TEACH
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Emory University (Other); Grady Health System (Other)
Responsible Party: Principal Investigator, Jeffrey Samet, Chief of General Internal Medicine, Boston Medical Center
Other Study IDs: H-33343; R01DA037768 (NIH)
Record Dates: First submitted 2015-08-12; First posted 2015-08-17 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: HIV Infection; Pain; Drug Dependence
Keywords: HIV Infection; Pain; Chronic Opioid Therapy; Addiction; Analgesics, Opioid
MeSH Terms: conditions — HIV Infections; Pain; Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Cohort: The TEACH patient cohort component will establish an observational cohort of HIV-infected patients on chronic opioid therapy.

SUMMARY:
The TEACH patient cohort will characterize a clinic sample of HIV-infected patients on chronic opioid therapy (COT) by describing basic demographics and health status, including characteristics of pain (severity and interference), aberrant behaviors/misuse of COT, substance use and trust/satisfaction with providers. In addition, data on a subset of participants will be used to supplement analysis of secondary outcomes for the TEACH randomized controlled trial (RCT), an intervention study directed at COT providers (outlined in a separate Clinical Trials Protocol Registration and Results (PRS) summary).

DETAILED DESCRIPTION:
The TEACH patient cohort study is multi-site and will be conducted at Boston Medical Center and Grady Memorial Hospital. It will involve recruiting and consenting HIV-infected patients on chronic opioid therapy (COT) to be participants in an observational study. The patient cohort will characterize a clinic sample of HIV-infected patients on COT by describing basic demographics and health status, including characteristics of pain (severity and interference), aberrant behaviors/misuse of COT, substance use and trust/satisfaction with providers. Participation in the study will involve completing one baseline and one follow-up assessment. The follow-up assessment will take place approximately 12 months after the baseline assessment. Both the baseline and follow-up assessments will be conducted at the clinical site, and a single signed consent form will be obtained for both visits. A similar assessment instrument will be used at baseline and follow-up. Additional health information will be collected from the medical record.

There are two distinct components to the TEACH study. The patient cohort component, which is outlined in this Clinical Trials PRS summary, will involve recruiting and consenting patients in the HIV clinic on COT to be participants in an observational study. The intervention, outlined in a separate Clinical Trials PRS summary, will involve consenting physicians as participants in a randomized controlled trial of an intervention and, via a waiver of informed consent, extracting patient level data on the physicians' patients from the electronic medical record. Data on a subset of observational cohort participants will be used to supplement analysis of secondary outcomes for the intervention (i.e. those patients whose providers were enrolled).

The TEACH patient cohort component seeks to inform physicians and other providers about patients who use chronic opioid therapy, including valuable information on the effect of the COT prescriber-directed intervention on patients. This knowledge will guide both prescribers and patients in improving care and reducing risks associated with chronic opioid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is HIV-infected
* Patient receives care in the HIV clinic at participating sites
* Patient is on chronic opioid therapy (e.g. 3 or more opioid prescriptions written at least 21 days apart in the prior 6 months)
* Patient is at least 18 years of age
* Patient can provide contact information for at least two contacts to assist with follow-up
* Patient has a home or mobile telephone
* Patient speaks English

Exclusion Criteria:

* Patient plans to move from area within 12 months
* Patient is unable to consent or understand interview (determined by trained research staff)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected COT patients from the HIV clinics at Boston Medical Center and Grady Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Pain severity in the past week (Brief Pain Inventory) | Participants will be followed up to one year
Opioid misuse (Current Opioid Misuse Measure) | Participants will be followed up to one year

SECONDARY OUTCOMES:
Pain interference in the past week (Brief Pain Inventory) | Participants will be followed up to one year
Any emergency department visit to seek opioids (medical chart review and interview) | Participants will be followed up to one year
Number of days of drug use in the past 30 days (Addiction Severity Index) | Participants will be followed up to one year
Trust in provider (Physician Trust Scale) | Participants will be followed up to one year
Satisfaction with COT (questions created) | Participants will be followed up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Samet, MD, MA, MPH, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.

REFERENCES:
- [Derived] Ngo B, Liebschutz JM, Cheng DM, Colasanti JA, Merlin JS, Armstrong WS, Forman LS, Lira MC, Samet JH, Del Rio C, Tsui JI. Hazardous alcohol use is associated with greater pain interference and prescription opioid misuse among persons living with HIV and chronic pain. BMC Public Health. 2021 Mar 22;21(1):564. doi: 10.1186/s12889-021-10566-6. PMID 33752634
- [Derived] Lira MC, Tsui JI, Liebschutz JM, Colasanti J, Root C, Cheng DM, Walley AY, Sullivan M, Shanahan C, O'Connor K, Abrams C, Forman LS, Chaisson C, Bridden C, Podolsky MC, Outlaw K, Harris CE, Armstrong WS, Del Rio C, Samet JH. Study protocol for the targeting effective analgesia in clinics for HIV (TEACH) study - a cluster randomized controlled trial and parallel cohort to increase guideline concordant care for long-term opioid therapy among people living with HIV. HIV Res Clin Pract. 2019 Apr;20(2):48-63. doi: 10.1080/15284336.2019.1627509. PMID 31303143